CLINICAL TRIAL: NCT04537780
Title: Clinical Study Evaluating the Efficacy and Safety of Montelukast in the Treatment of Non-Alcoholic Steatohepatitis (NASH)
Brief Title: Efficacy and Safety of Montelukast in Non Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dr. Tarek Mohamed Mostafa, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Montelukast
Record Dates: First submitted 2020-08-30; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: randomized, prospective placebo controlled study that will be conducted on 44 patients who fulfill the selection criteria and will be classified randomly into two groups.
  Group 1 (Control group n= 22): Patients will receive Placebo once daily at bedtime.
  Group 2 (Treatment group n= 22): Patients will receive Montelukast 10 mg daily at bedtime. The treatment duration will be 12 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Placebo Comparator): (Control group n= 22): Patients will receive Placebo once daily at bedtime for 12 weeks..
  Interventions: Other: Placebo
- Group 2 (Experimental): Treatment group n= 22): Patients will receive Montelukast 10 mg daily at bedtime.
  The treatment duration will be 12 weeks.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Other: Placebo — Placebo tabled every day
  Arms: group 1
Drug: Montelukast — Montelukast 10 mg daily at bed time.
  Other Names: Singulair
  Arms: Group 2

SUMMARY:
the current study is to evaluate the efficacy and safety of Montelukast in the treatment of patients with non-alcoholic steatohepatitis (NASH).

DETAILED DESCRIPTION:
This is a randomized, prospective placebo-controlled study that will be conducted on 44 patients who fulfill the selection criteria and will be classified randomly into two groups.

Group 1 (Control group n= 22): Patients will receive Placebo once daily at bedtime.

Group 2 (Treatment group n= 22): Patients will receive Montelukast 10 mg daily at bedtime.

The treatment duration will be 12 weeks. Patients will be recruited from National Liver Institute and Fever, Liver and GIT disease Shebin El-Kom hospital, Egypt. All participants will be informed about the nature of the study. The patients will give their informed consent.The study will be approved by Research Ethics Committee of faculty of pharmacy -Tanta University. Data of all patients will be private and confidential. Any unexpected risk will be reported to patients and ethical committee on time

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) overweight/obese subjects who have persistently abnormal aminotransferase level in two separate occasions over the past six months.

NAFLD will be assumed in patients with moderately elevated aminotransferase activities (<3x the upper limit of normal).

There is evidence of hepatic steatosis by imaging (increased liver echogenicity (bright), stronger echoes in the hepatic parenchyma, vessel blurring, and narrowing of the lumen of the hepatic veins) and there is no cause for secondary hepatic fat accumulation such as significant alcohol consumption, use of steatogenic medication or hereditary disorders. Patients with fibroscan score >7 kPa and <14 kPa will be included in the study.

Exclusion Criteria:

* Alcohol abusers.
* Presence of evidence for viral or autoimmune hepatitis.
* Diabetic patients.
* Patients with Wilson's disease and patients with hemochromatosis.
* Patients with decompensated liver disease.
* Patients show hypersensitivity to studied medications.
* Patients taking medication known to cause steatosis.
* Patients with other comorbid conditions that could potentially elevate transaminase, such as congestive heart failure, malignancy.
* Pregnancy and lactating women.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
serum 8-Hydroxy2-deoxyguanisine (8-OHdG) | 12 Weeks
  Quantitative detection of human 8-OHdG will be done using commercially available Enzyme-linked Immunosorbent assay kits.
TNF-α. | 12 Weeks
  Quantitative detection of TNF-α will be done using commercially available Enzyme-linked Immunosorbent assay kits.
Alanine aminotransferase (ALT). | 12 Weeks
  ALT will be measured by colorimetric method.
Aspartate aminotransferase (AST) | 12 Weeks
  AST will be measured by colorimetric method.
ɤ-glutamyltranspeptidase(GGT) | 12 Weeks
  ɤ-glutamyltranspeptidase(GGT) will be measured by colorimetric method.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Mostafa, Ass. Prof., Study Director — Tanta University
Locations (1):
- Dr. Tarek Mohamed Mostafa, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Said MM, Bosland MC. The anti-inflammatory effect of montelukast, a cysteinyl leukotriene receptor-1 antagonist, against estradiol-induced nonbacterial inflammation in the rat prostate. Naunyn Schmiedebergs Arch Pharmacol. 2017 Feb;390(2):197-205. doi: 10.1007/s00210-016-1325-4. Epub 2016 Dec 1. PMID 27909742
- [Background] Kuru S, Kismet K, Barlas AM, Tuncal S, Celepli P, Surer H, Ogus E, Ertas E. The Effect of Montelukast on Liver Damage in an Experimental Obstructive Jaundice Model. Viszeralmedizin. 2015 Apr;31(2):131-8. doi: 10.1159/000375434. Epub 2015 Apr 9. PMID 26989383